CLINICAL TRIAL: NCT04030793
Title: Individualized Transcranial Direct Current Stimulation for Gait Function in Healthy Subjects
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated due to difficulty in recruiting subjects
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2018-11-021
Record Dates: First submitted 2019-07-21; First posted 2019-07-24 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Healthy Adults; Healthy Aging
Keywords: Brain Stimulation; Transcranial direct current stimulation; Motor function

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized stimulation group (Experimental): Based on transcranial direct current stimulation (tDCS) simulation, individualized stimulation on leg motor areas during 30 minutes.
  Interventions: Device: Individualized transcranial direct current stimulation
- Conventional stimulation group (Active Comparator): Conventional stimulation on leg motor areas during 30 minutes.
  Interventions: Device: Conventional transcranial direct current stimulation

INTERVENTIONS:
Device: Individualized transcranial direct current stimulation — Based on tDCS stimulation, individualized stimulation during 30 minutes with sitting position.
  Arms: Individualized stimulation group
Device: Conventional transcranial direct current stimulation — Conventional tDCS stimulation during 30 minutes with sitting position.
  Arms: Conventional stimulation group

SUMMARY:
The purpose of this study is to compare the effects of individualized brain stimulation based on simulation and conventional brain stimulation in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

• Healthy adult men and women without history of central nervous system disease and abnormalities

Exclusion Criteria:

* Under 18 years old, 75 years old or older
* A person who has inserted a metal object in a skull
* A person with complete occlusion of the carotid artery
* A person with epilepsy
* Pregnant and lactating women
* Who is not eligible for the test

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-08-29 (Actual)

PRIMARY OUTCOMES:
Changes in cortical activation | Change from baseline (before stimulation) after stimulation during 30 min
  changes in cortical activation is measured by functional Near-Infrared-Spectroscopy (fNIRS) (NIRScout, NIRx, Germany) during treadmill gait.

SECONDARY OUTCOMES:
10 meter walk test (10MWT) | Before stimulation (baseline); After strimulation during 30 min
  Measure of self selected speeds by measuring the time it takes an individual to walk 10 meters. To perform the test, patient walks 10 meters (33 ft) and the time is measured when the leading foot crosses the start line and the finish line. The instructions are: "Please walk this distance at your normal pace when I say go."
Timed Up and Go test (TUG) | Before stimulation (baseline); After strimulation during 30 min
  The Timed Up and Go test (TUG) is a simple test used to assess a person's mobility and requires both static and dynamic balance. It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down.
Gait analysis using surface electromyograph | Before stimulation (baseline); After strimulation during 30 min
  Gait analysis is a process of measuring and evaluating the walking patterns of patients by using surface electromyograph.
Gait analysis using motion analysis system | Before stimulation (baseline); After strimulation during 30 min
  Gait analysis is a process of measuring and evaluating the walking patterns of patients by using motion analysis system.

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Hee Kim, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided